CLINICAL TRIAL: NCT05552950
Title: Randomized, Controlled, Double-Blind Proof of Concept Trial Assessing the Efficacy and Safety of BioBlock® Intranasally Administered Virus-Neutralizing Bovine Colostrum Nasal Spray in Preventing of COVID-19 Infection in Healthy Volunteer Individuals
Brief Title: The Efficacy and Safety of BioBlock® Intranasally Administered Virus-Neutralizing Bovine Colostrum Nasal Spray in Preventing of COVID-19 (Coronavirus Disease-19) Infection in Healthy Volunteer Individuals
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chemi-Pharm AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BioBlock
Record Dates: First submitted 2022-09-09; First posted 2022-09-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-09

CONDITIONS: SARS CoV 2 Infection
Keywords: SARS-CoV-2; COVID-19; nasal spray; Antiviral agent
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The study and control sprays can only be distinguished by serial numbers, the content of which is not known by the study staff or the subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Individuals using the BioBlock® antiviral nasal spray immediately after waking up in the morning and thereafter once every 4 hours and so for 28 days.
  Interventions: Biological: BioBlock® antiviral nasal spray
- control group (Placebo Comparator): Placebo is used by individuals immediately after waking up in the morning and thereafter once every 4 hours and so for 28 days.
  Interventions: Biological: BioBlock® antiviral nasal spray

INTERVENTIONS:
Biological: BioBlock® antiviral nasal spray — SARS-CoV-2 BioBlock is a natural preparation derived from bovine colostrum, where animals have an immune response against the SARS-CoV-2 spike protein in addition to conventional vaccines. The antiviral colostrum preparation was made from colostrum of cows immunized with SARS CoV-2 spike protein. Pregnant cows were immunized during the third trimester of gestation using a non-infectious recombinantly produced and purified SARS CoV-2 spike protein. Colostrum, which is milked after calving, concentrates most of the antibodies produced in the cow's body at very high concentrations, including neutralizing antibodies to SARS CoV-2 produced as a result of immunization.

SUMMARY:
This is a proof-of-concept double-blind cluster randomized (1:1) parallel study. The randomization unit is healthy volunteers who have no symptoms of COVID-19 at the start of the study and have not been infected with the SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2) virus in the past 90 days. The selected individuals are randomly grouped in either the experimental group (individuals using the BioBlock® antiviral nasal spray immediately after waking up in the morning and thereafter once every 4 hours and so for 28 days) or the control group (placebo is used by individuals immediately after waking up in the morning and thereafter once every 4 hours and so for 28 days).

ELIGIBILITY:
Inclusion Criteria:

Agree to participate in the study Age: 18-60 years (based on the age group with the best digital competence).

Exclusion Criteria:

* Pregnancy
* age less than 18 years and over 60 years,
* a person identified with SARS-CoV-2 infection at the beginning of the study,
* a person with symptoms of SARS-CoV-2 infection,
* a person who has recovered from Covid-19 in the last 3 months,
* a person who regularly takes medicinal products administered by inhalation by nasal and oropharyngeal means.
* patients with known allergies to BioBlock® components and milk proteins

  * BioBlock ingredients are: Purified water • Bovine colostrum SARS-CoV-2 antibodies • Phosphate buffer: DPBS (without Ca and Mg salts) • Viscosity-enhancing agents: PEG400, PVP K30 • Preservative: sodium benzoate • Acidity regulator: citric acid • Mucous membrane moisturizing agent: glycerol • Potassium chloride - buffer solution component • Potassium dihydrogen phosphate - buffer solution component • Sodium chloride - buffer solution component • Disodium phosphate - buffer solution component
  * .
* BioBlock® use in the last 24 hours If the subject has taken BioBlock® during the last day and there are no other criteria for exclusion from the study, then the subject is suitable for inclusion in the study from the next day

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2000 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
effectiveness of the BioBlock® | 3 months
  BioBlock® nasal spray users are less likely to contract the virus than placebo users. BioBlock effectiveness will be estimated using Cox regression (BPE = 1 - hazard ratio [HR]) or Poisson regression (BPE = 1 - rate ratio [RR]).

SECONDARY OUTCOMES:
safety of the BioBlock® virus neutralizing nasal spray | 6 months
  The use of BioBlock® nasal spray does not cause life-threatening or other significant side effects. Incidence of all possible side effects that person or medical person connects to the use of the product. Side effects are not pre-specified because of the nature of product. Number (%) of adverse events per group are reported. Mean (sd) and median (IQR) duration of symptoms is calculated and compared between groups using linear regression with cluster robust standard errors in case of correlated observations or t-test or Wilcoxon rank-sum test.

CONTACTS AND LOCATIONS:
Locations (1):
- AS Chemi-Pharm, Tallinn, Harju, Estonia

IPD SHARING:
Plan to Share IPD: Undecided